CLINICAL TRIAL: NCT06042075
Title: Representation of Congenital Birthmarks in Newborns by Angers Maternity Unit Health Professionals
Brief Title: Representation of Congenital Birthmarks
Acronym: ReCONNAISSANCE
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2023-0-100
Record Dates: First submitted 2023-09-11; First posted 2023-09-18 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: Body Representation; Congenital Skin Disorder; Feelings
Keywords: Newborns; Health Professionals; Maternity Unit; Congenital Birthmarks
MeSH Terms: conditions — Skin Abnormalities

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Health professionals: Health professionals working at Angers Maternity Unit include gynecologists, pediatricians, residents (gynecology and pediatric residents), childcare assistants, nursing auxiliaries and midwives.
  Interventions: Other: Questionnaire on congenital birthmarks

INTERVENTIONS:
Other: Questionnaire on congenital birthmarks — Questions will be put to health professionals on representation using a semi-quantitative questionnaire.

SUMMARY:
This descriptive cross-sectional single center study will be conducted at Angers Maternity Unit.

It pertains to the ways in which healthcare professionals represent congenital birthmarks found in newborns.

It is our assumption that health professionals may have a tendency to engage in inappropriate behavior when dealing with congenital birthmarks due to lack of knowledge. We make the presumption that insufficient knowledge causes difficulties in managing these birthmarks.

Data as to representation of birthmarks in newborns by health professionals will be collected using a semi-quantitative questionnaire.

This study constitutes preliminary research work, with a view to creating a professional development plan if necessary.

DETAILED DESCRIPTION:
This descriptive cross-sectional observational study will take place at a single center: Angers Hospital Maternity Unit.

Our aim is to assess how healthcare professionals represent congenital birthmarks in newborn infants.

We intend to use an optional anonymous questionnaire that will be placed strategically in Angers Maternity Unit workspaces . Each health professional from Angers Maternity Unit will be asked to complete this questionnaire.

In this five-minute questionnaire, they will be asked questions regarding their representation of congenital birthmarks, their feelings and their knowledge.

We make the hypothesis that some health professionals lack knowledge and are uncomfortable with managing these birthmarks and providing explanations to the parents of newborn infants. We also show them some examples of birthmarks, prompting them to express any feelings they may have.

This questionnaire was co-written by Pauline VABRES, a psychologist with experience in the field of self-representation.

The questionnaire will remain accessible for 45 days, ensuring that every Maternity Unit health professional has the opportunity to participate (approximately 140 people, excluding non-health professionals working in the Maternity Unit and students).

On completion of the questionnaire, the healthcare professionals will seal their answers in envelopes to guarantee anonymity.

At the end of the 45-day period, the answers will be collected and analyzed.

If required, the second phase of this work will focus on developing educational interventions for health professionals to enhance their knowledge of congenital birthmarks. We also hope to improve management of these lesions and enhance the quality of the explanations provided to parents of newborns.

Previous studies have already addressed the feelings of parents confronted with congenital birthmarks. To our knowledge, this is the first study of its kind to evaluate the perspective of health professionals

ELIGIBILITY:
Inclusion Criteria

All health professionnals working at Angers Maternity Unit:

* Midwives
* Nursing auxiliaries
* Childcare assistants
* Gynecologists
* Residents
* Pediatricians

Exclusion Criteria:

* Refusal to participate
* Non-health professionals working at Angers Maternity Unit (hospital cleaners, hospital food workers)
* Students (trainee pediatricians, trainee gynecologists, trainee midwives)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All health professionnals working at Angers Maternity Unit: midwives, nursing auxiliaries, childcare assistants, gynecologists, residents, pediatricians
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2023-11 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Assessment of the ways in which health professionals from Angers Maternity Unit represent congenital birthmarks found in newborns | 45 days
  Representation by health professionals will be assessed using a semi-quantitative questionnaire

SECONDARY OUTCOMES:
Assessment of the proportion of health professionals wishing to improve their knowledge of congenital birthmarks | 45 days
  The question will be put to health professionals using a questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Dermatology, University Hospital of Angers, Angers, Pays de Loire, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kelly KA, Balogh EA, Kaplan SG, Feldman SR. Skin Disease in Children: Effects on Quality of Life, Stigmatization, Bullying, and Suicide Risk in Pediatric Acne, Atopic Dermatitis, and Psoriasis Patients. Children (Basel). 2021 Nov 16;8(11):1057. doi: 10.3390/children8111057. PMID 34828770
- [Background] Vivar KL, Kruse L. The impact of pediatric skin disease on self-esteem. Int J Womens Dermatol. 2017 Dec 12;4(1):27-31. doi: 10.1016/j.ijwd.2017.11.002. eCollection 2018 Mar. PMID 29872673
- See also: Effects on Quality of Life, Stigmatization, Bullying, and Suicide Risk in Pediatric Acne, Atopic Dermatitis, and Psoriasis Patients — https://pubmed.ncbi.nlm.nih.gov/29872673/
- See also: The impact of pediatric skin disease on self-esteem — https://pubmed.ncbi.nlm.nih.gov/34828770/